CLINICAL TRIAL: NCT05305482
Title: Drug-Coated Stent Versus Drug-Eluting Stent for One-month Dual-antiplatelet Therapy in Patients With Acute Coronary Syndrome: ONE-PASS Trial
Brief Title: DCS Versus DES for One-month DAPT in Patients With ACS: ONE-PASS Trial
Acronym: ONE-PASS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Chul-Min Ahn, Professor, Principal Investigator, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-2021-0089
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; Drug-eluting stent; Dual-antiplatelet therapy; Ticagrelor
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Drug-Eluting Stents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DCS group (Experimental): Drug-coated stent group
  Interventions: Device: Drug-coated stent
- DES group (Active Comparator): Drug-eluting stent group
  Interventions: Device: Drug-eluting stent

INTERVENTIONS:
Device: Drug-coated stent — The polymer-free drug-coated stent (BioFreedom Ultra stent) will be implanted for the DCS group.
  Other Names: BioFreedom Ultra stent
  Arms: DCS group
Device: Drug-eluting stent — The Biodegradable polymer drug-eluting stent (Ultimaster stent) will be implanted for the DES group.
  Other Names: Ultimaster stent
  Arms: DES group

SUMMARY:
To test whether the polymer-free drug-coated stent (DCS) BioFreedom is noninferior to the biodegradable polymer drug-eluting stent (DES) Ultimaster in terms of 1-year patient-oriented composite endpoint (POCE, composite of all-cause mortality, any MI, or any revascularization) in a setting of 1-month dual-antiplatelet therapy (DAPT) strategy (1-month DAPT followed ticagrelor monotherapy) after acute coronary syndrome.

DETAILED DESCRIPTION:
This trial is an open-label, randomized, multi-center study. Patients with ACS requiring percutaneous coronary intervention will be randomized with a 1:1 ratio either of DCS group or DES group. After the index procedure, DAPT (100 mg aspirin qd and 90 mg ticagrelor bid) will be given for 1 month. After this, ticagrelor monotherapy will be maintained for 11 months. Clinical events will be evaluated within 12 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥19 years
2. All subjects who are acceptable candidates for treatment with a drug-coated stent or drug-eluting stent because of acute coronary syndrome
3. Provision of informed consent

Exclusion Criteria:

1. Current or potential pregnancy
2. Need of oral anticoagulation therapy
3. Inability to follow the patient over the period of 1 year after enrollment, as assessed by the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3520 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2030-02-14 (Estimated); Study Completion 2030-02-14 (Estimated)

PRIMARY OUTCOMES:
Patient-Oriented Composite Endpoint (POCE) | At 1 year after randomization
  The composite of all-cause death, MI, or any revascularization

SECONDARY OUTCOMES:
Device-Oriented Composite Endpoint (DOCE) | At 1 year after randomization
  The composite of cardiovascular death, MI (not clearly attributable to a non-target vessel), or clinically-driven target-lesion revascularization (TLR)
All-cause death | At 1 year after randomization
  All death including cardiovascular death
Cardiovascular death | At 1 year after randomization
  Death resulting from cardiovascular causes or undetermined cause of death not attributable to any other category because of the absence of any relevant source documents
Myocardial infarction | At 1 year after randomization
  A spontaneous event according to the fourth universal definition of myocardial infarction and the Academic Research Consortium-2 Consensus Document
Stroke | At 1 year after randomization
  Loss of neurologic function caused by an ischemic or hemorrhagic event
Stent thrombosis (definite or probable) | At 1 year after randomization
  By the Academic Research Consortium-2 Consensus Document
Any revascularization | At 1 year after randomization
  All revascularizations including target-vessel revascularization and and non-target-vessel revascularization
Target-vessel revascularization | At 1 year after randomization
  Clinically indicated or ischemia driven any repeat percutaneous intervention or surgical bypass of any segment of the target vessel including the target lesion
Non-target vessel revascularization | At 1 year after randomization
  Clinically indicated or ischemia driven any repeat percutaneous intervention or surgical bypass of any segment of the non-target vessel
Target-lesion revascularization | At 1 year after randomization
  Clinically indicated or ischemia driven repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion
BARC type 2-5 bleeding | At 1 year after randomization
  According to a consensus report from the Bleeding Academic Research Consortium
BARC type 3-5 bleeding | At 1 year after randomization
  According to a consensus report from the Bleeding Academic Research Consortium

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Min Ahn, Principal Investigator — Yonsei University Health System, Severance Hospital
Locations (1):
- Yonsei Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
The data will be available from the principal investigator on reasonable request.